CLINICAL TRIAL: NCT03019107
Title: Breath Synchronized Abdominal Muscle Stimulation to Facilitate Ventilator Weaning: a Pilot
Brief Title: Breath Synchronized Abdominal Muscle Stimulation to Facilitate Ventilator Weaning: a Pilot Study
Status: Terminated | Type: Interventional
Why Stopped: Unable to meet enrollment goal
Sponsor: Liberate Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LM-KINDRED-01
Record Dates: First submitted 2016-12-13; First posted 2017-01-12 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Electric Stimulation; Respiration, Artificial; Ventilator Weaning
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- VentFree Stimulation (Experimental): Breath synchronized abdominal NMES
  Interventions: Device: Breath synchronized abdominal NMES
- Sham Stimulation (Sham Comparator): Sham breath synchronized abdominal NMES
  Interventions: Device: Sham breath synchronized abdominal NMES

INTERVENTIONS:
Device: Breath synchronized abdominal NMES — VentFree prototype (VF03) that delivers electrical stimulation pulses to the abdominal muscles during exhalation with a frequency of 30 Hz, a pulse width of 350 µs and 90% of the maximum current that the participant can tolerate. These stimulation parameters were selected to cause a tetanic (continuous) contraction of the abdominal muscles, without pain for the patient. Stimulation will be administered for 30 minutes 2 times per day, 5 days per week, for 6 weeks; or until the patient is weaned from mechanical ventilation.
  Other Names: VentFree
  Arms: VentFree Stimulation
Device: Sham breath synchronized abdominal NMES — Modified VentFree prototype (VF03) that delivers stimulation pulses to the abdominal muscles during exhalation with a frequency of 10 Hz, a pulse width of 100 µs and current set to 10 milliamp. These stimulation parameters were chosen to cause a twitch contraction of the abdominal wall muscles. Stimulation will be administered for 30 minutes, 2 times per day, 5 days per week, for 6 weeks; or until the patient is weaned from mechanical ventilation.
  Arms: Sham Stimulation

SUMMARY:
The primary objective of this study is to determine whether neuromuscular electrical stimulation applied to the abdominal wall muscles in synchrony with exhalation can increase the strength of the respiratory muscles in prolonged mechanical ventilation patients.

DETAILED DESCRIPTION:
In the U.S. over 500,000 patients have difficulty weaning from mechanical ventilation every year. These patients cost the health care system $16 billion annually and have an increased risk of medical complications and morbidity.

A major factor responsible for weaning failure is the imbalance between decreased respiratory muscle strength and excessive respiratory load. This study includes an investigational device that applies electrical stimulation to the abdominal muscles in synchrony with exhalation. This is hypothesized to improve the strength of the respiratory muscles. The long term goal of this project is to determine whether this approach can reduce the number of days taken for patients to wean from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been mechanically ventilated for at least fourteen days.
* Clinically stable: oxygen saturation > 90% with a fractional inspired oxygen ≤ 0.40, external positive end expiratory pressure ≤ 5 centimeters water, temperature ranging from 35.5 to 38.5 degrees celsius, no intravenous administration of vasoactive agents.

Exclusion Criteria:

* Patients in whom Neuromuscular Electrical Stimulation (NMES) does not elicit a palpable contraction of the abdominal muscles.
* Patients with broken or irritated skin on the abdominal wall
* Patients with a history of neuromuscular disease
* Body Mass Index (BMI) > 35 kg/m2
* Patients who are not medically stable
* Patients with a pacemaker
* Female patients who are pregnant
* Patients under the age of 18
* Patients who are expected to die within four weeks
* Patients who are unable to follow verbal instructions
* Patients with epilepsy
* Patients with an abdominal wall hernia
* Patients with anoxic encephalopathy
* Patients with history of, or active, substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kindred Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VentFree Stimulation | Sham Stimulation
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the control group as the trial was terminated after the first patient was enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | VentFree Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Duration of mechanical ventilation at enrollment [Number; unit: Days] | 18 |  | 18
Primary reason for mechanical ventilation [Count of Participants; unit: Participants]
  Acute Respiratory Failure | 1 |  | 1
  Coma | 0 |  | 0
  COPD | 0 |  | 0
  Asthma | 0 |  | 0
  Neuromuscular Disease | 0 |  | 0
Cause of acute respiratory failure [Count of Participants; unit: Participants]
  Pneumonia | 1 |  | 1
  Other | 0 |  | 0
Acute Physiology and Chronic Health Evaluation II (APACHE II) score [Number; unit: units on a scale] — The APACHE II score is a widely used ICU prognostic scale that is a measurement of patient disease severity and strongly correlates with patient outcomes.
  The APACHE II is an integer score from 0 to 71; higher scores correspond to more severe disease and a higher risk of death.
  units on a scale | 13 |  | 13
Tracheostomized [Count of Participants; unit: Participants]
  Tracheostomized | 1 |  | 1
  Not Tracheostomized | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Expiratory Pressure From Baseline to Extubation
Description: Maximum expiratory pressure was measured from total lung capacity
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: No patients were enrolled in the sham arm
Measure: Number; unit: cmH2O
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
cmH2O | 2 |

2. Primary Outcome: Change in Maximum Inspiratory Pressure From Baseline to Extubation
Description: Maximum inspiratory pressure was measured from end expiratory lung volume.
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: No patients were enrolled in the sham arm
Measure: Number; unit: cmH2O
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
cmH2O | 8 |

3. Secondary Outcome: Change in Thickness of the Transverse Abdominis Muscle From Baseline to Extubation
Description: Thickness of transverse abdominis muscle as measured by ultrasound
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: This measurement was not collected due to equipment problems.
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Thickness of the External Oblique Muscle From Baseline to Extubation
Description: Thickness of the external oblique muscle as measured by ultrasound
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: This measurement was not collected due to equipment problems.
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Thickness of the Internal Oblique Muscle From Baseline to Extubation
Description: Thickness of the internal oblique muscle as measured by ultrasound
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: This measurement was not collected due to equipment problems.
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Thickness of the Rectus Abdominis Muscle
Description: Thickness of the rectus abdominis muscle as measured by ultrasound
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: This measurement was not collected due to equipment problems.
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Thickness of the Diaphragm
Description: Thickness of the diaphragm as measured by ultrasound
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: This measurement was not collected due to equipment problems.
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Weaning Success
Description: Defined as free from ventilator support for more than 72 hours
Time Frame: The earlier of 6 weeks or first extubation, an expected average of 4 weeks
Population: No participants were enrolled in the sham group
Measure: Count of Participants; unit: Participants
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
Participants | 0 |

9. Secondary Outcome: Number of Days Taken to Wean
Time Frame: The earlier of 6 weeks or first extubation, an expected average of 4 weeks
Population: No patients in the treatment group were successfully extubated from the ventilator. No patients were enrolled in the sham group
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Cough Peak Flow From Baseline to Extubation
Description: Cough peak flow was measured from total lung capacity
Time Frame: Change from baseline to first extubation, an expected average of 4 weeks
Population: No participants were enrolled in the sham group
Measure: Number; unit: Liters per minute
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
Liters per minute | 21 |

11. Secondary Outcome: Change in Spontaneous Tidal Volume From Baseline to Final Visit or First Extubation
Time Frame: Change from baseline to final study visit or first extubation, an expected average of 4 weeks
Population: No participants were enrolled in the sham stimulation group.
Measure: Number; unit: milliliters
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
milliliters | 150 |

12. Secondary Outcome: Change in Spontaneous Respiratory Rate From Baseline to Final Study Visit
Time Frame: Change from baseline to final study visit, an expected average of 4 weeks
Population: No participant were enrolled in the sham group
Measure: Number; unit: breaths per minute
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
breaths per minute | -5 |

13. Secondary Outcome: Change in Spontaneous Minute Ventilation From Baseline to Final Study Visit
Time Frame: Change from baseline to final study visit, an expected average of 4 weeks
Population: No participants were enrolled in the sham group
Measure: Number; unit: liters per minute
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
liters per minute | -1.2 |

14. Secondary Outcome: Maximum Sensation of Stimulation Experienced by Patient
Description: Measured using the behavioral pain scale
Time Frame: Through study completion, an expected average of 4 weeks
Population: This measurement was not recorded.
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Adverse Events That Are Related to Treatment
Description: This includes any adverse event that was graded as having a possible, probable or definite relationship to the study intervention.
Time Frame: Though study completion, an expected average of 4 weeks
Population: No participants enrolled in sham group
Measure: Number; unit: events
Arm/Group | VentFree Stimulation | Sham Stimulation
Number analyzed (Participants) | 1 | 0
events | 1 |

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse events were reviewed during every study intervention session
Arm/Group | VentFree Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VentFree Stimulation (N=1) | Sham Stimulation (N=0)
Mean arterial pressure (Cardiac disorders) | 1 (1) | NA — Mean arterial pressure was elevated to 128 mmHg prior to initiation of treatment. Adverse event was assessed with Moderate severity, no relationship with study device, and was resolved with no sequel.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Adverse event was assessed with Moderate severity and unrelated to study intervention. Resolved with no sequel.
Abdominal muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | NA — Adverse event was rated with Mild severity and Definitely related to study intervention. Resolved with no sequel

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03019107/Prot_SAP_001.pdf